CLINICAL TRIAL: NCT03714646
Title: The Effects of Beta Glucan on Acetate Production and Human Substrate Metabolism
Brief Title: Beta Glucan and Acetate Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL63759.068.17
Record Dates: First submitted 2018-07-06; First posted 2018-10-22 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2018-10

CONDITIONS: Pre Diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — beta-Glucans; Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- beta glucan (Active Comparator)
  Interventions: Dietary Supplement: beta gluten
- beta glucan and Resistant Starch (Experimental)
  Interventions: Dietary Supplement: beta glucan and resistant starch

INTERVENTIONS:
Dietary Supplement: beta glucan and resistant starch — 12g per day the day before the CID Resistant starch 7.5 g
  Arms: beta glucan and Resistant Starch
Dietary Supplement: Placebo — isocaloric maltodextrin before the CID
  Arms: Placebo
Dietary Supplement: beta gluten — 12 g beta gluten there day before the CID
  Arms: beta glucan

SUMMARY:
Based on our hypothesis that orally administered resistant starch and beta glucan will be fermented into a SCFA pattern high in acetate and that this will lead to beneficial effects on human substrate and energy metabolism, we aim to address the following primary objective:

To investigate the effects of an acute administration of inulin/beta glucan in combination with resistant starch on fecal and plasma acetate, as well as on fasting and postprandial substrate and energy metabolism in lean normoglycemic men and obese, prediabetic men.

ELIGIBILITY:
Inclusion Criteria:

* lean (BMI ≥ 20kg/m2 and ≤ 24.9kg/m2)
* normoglycemic
* aged 30 - 65 years

OR

* overweight/obese (BMI ≥ 25kg/m2 and ≤ 34.9kg/m2)
* pre-diabetes
* aged between 30 - 65 years.

Exclusion Criteria:

* diabetes mellitus
* gastroenterological diseases or major abdominal surgery (allowed i.e.: ---appendectomy, cholecystectomy)
* lactose intolerance and other digestive disorders
* cardiovascular disease, cancer, liver or kidney malfunction (determined based on ALAT and creatinine levels, respectively)
* disease with a life expectancy shorter than 5 years
* Use of antibiotics 3 months prior inclusion
* Use of probiotics or prebiotics

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Plasma acetate concentrations (microM) | at baseline (before a high-fat mixed meal)
Plasma acetate concentrations (microM) | four hours after a high fat mixed meal

SECONDARY OUTCOMES:
Energy expenditure (kJ/min) will be measured using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | at baseline and four hours after a high fat mixed meal
fat oxidation (g/min) will be measured using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | at baseline and four hours after a high fat mixed meal
carbohydrate oxidation (g/min) will be measured using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | at baseline and four hours after a high fat mixed meal
Circulating hormone concentrations (Insulin, GLP-1, PYY) | at baseline and four hours after a high fat mixed meal
Circulating metabolite concentrations (Glucose, Free Fatty Acids, Triglycerides) | at baseline and four hours after a high fat mixed meal
Plasma glucose (mmol/L) | at baseline and four hours after a high fat mixed meal
Free Fatty Acids (micromol/L) | at baseline and four hours after a high fat mixed meal
Breath H2 using (Bedfont EC60 Gastrolyzer, Rochester, UK) | at baseline and four hours after a high fat mixed meal

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Canfora EE, Hermes GDA, Muller M, Bastings J, Vaughan EE, van Den Berg MA, Holst JJ, Venema K, Zoetendal EG, Blaak EE. Fiber mixture-specific effect on distal colonic fermentation and metabolic health in lean but not in prediabetic men. Gut Microbes. 2022 Jan-Dec;14(1):2009297. doi: 10.1080/19490976.2021.2009297. PMID 34923911